CLINICAL TRIAL: NCT04980326
Title: A Scalable Low-intensity Psychological Intervention to Reduce Psychological Distress Among Healthcare Workers Involved in the First COVID-19 Outbreak in Spain: a Randomized Trial
Brief Title: A Scalable Psychological Intervention to Reduce Psychological Distress Among Healthcare Workers
Acronym: RESPOND-HCW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Universidad Autonoma de Madrid (Other); Hospital Universitario La Paz (Other); Parc Sanitari Sant Joan de Déu (Other); Fundació Sant Joan de Déu (Other); European Commission (Other); VU University of Amsterdam (Other); World Health Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RESPOND WP4 RCT
Record Dates: First submitted 2021-07-16; First posted 2021-07-28 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2021-11

CONDITIONS: Psychological Distress; Depression; Anxiety
Keywords: COVID-19; Healthcare workers; Psychological Distress; Depression; Anxiety; Problem Management Plus (PM+); Doing What Matters (DWM); Stepped-care
MeSH Terms: conditions — Depression; Anxiety Disorders; COVID-19 | interventions — Psychological First Aid

STUDY DESIGN:
Intervention Model Description: Participants will be allocated to the experimental or the control arm with a 1:1 ratio. Participants in the experimental arm will first received the step 1 of the stepped-care program, namely the Doing What Matters self-guided program. If they still report significant levels of psychological distress, as measured by the K-10 scale, 1 week after DWM, they will be invited to step 2, an individual intervention namely Problem Management Plus (PM+). If they do not report significant levels of psychological distress, they will not receive further interventions, but will be asked to complete the remaining assessments.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will not know whether a single participant was allocated to the experimental or to the control arm. That will be done by assigning random values toe the variable "arm" in the dataset.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stepped-care program (Step 1: DWM; Step 2: PM+) (Experimental): The treatment group will receive the stepped-care program consisting of Doing What Matters (DWM) (step 1) and Problem Management Plus (PM+) (step 2) in addition to Psychological First Aid (PFA) and care-as-usual (CAU). Step 2 will only be provided if the participant still has elevated levels of psychological distress at 2 weeks after DWM, i.e. during the second quantitative assessment at 2 weeks after DWM.
  Participants allocated to the experimental arm will also receive training in PFA, which consists of a 30-min call that covers basic aspects about peer support in times of stress. Participants will also be allowed to continue with their mental health interventions (CAU), as long as they meet eligibility criteria.
  Interventions: Behavioral: Doing What Matters (DWM); Behavioral: Problem Management Plus (PM+); Behavioral: Psychological First Aid (PFA)
- Psychological First Aid (PFA) (Active Comparator): Participants allocated to the control arm will also receive training in PFA, which consists of a 30-min call that covers basic aspects about peer support in times of stress. Participants will also be allowed to continue with their mental health interventions (CAU), as long as they meet eligibility criteria.
  Interventions: Behavioral: Psychological First Aid (PFA)

INTERVENTIONS:
Behavioral: Doing What Matters (DWM) — The original DWM program consists of a self-help guide called 'Doing What Matters in Times of Stress', that is complemented with pre-recorded audio exercises. The audio material imparts key information about stress management and guides participants through individual exercises. Additionally, participants are guided by a briefly trained helper. In this study, DWM will be delivered as an online intervention. The DWM intervention, i.e. both the audio recordings and the self-help guide, will be adapted for use on a smartphone or other device with internet access during Phase 1 of RESPOND. The format of DWM is innovative in that it seeks to ensure that key intervention components are delivered as intended through the use of pre-recorded audio, without the burden of extensive training and supervision. In the online application tool a new module is released every week so participants will be asked to go through the entire DWM intervention within 5 weeks with weekly guidance from a helper.
  Other Names: Doing What Matters in Times of Stress; Self Help Plus; SH+; DWM
  Arms: Stepped-care program (Step 1: DWM; Step 2: PM+)
Behavioral: Problem Management Plus (PM+) — PM+ is a new, brief, psychological intervention program based on cognitive behavioral therapy (CBT) techniques. The manual involves the following empirically supported elements: problem solving plus stress management, behavioral activation, facing fears, and accessing social support. Across the five 90-minute sessions participants may talk to trained non-professional. PM+ has four core features, and it is brief. In this study, the delivery mode of the PM+ intervention will be flexible, with remote delivery in phases of the pandemic when physical distancing rules apply. This is a future-oriented attempt towards a more holistic mental health care system that can flexibly switch between modes of delivery (e.g. remotely (e.g. Zoom) or face-to), depending on the needs and the specific containment measures that apply, and the specific preferences and needs of the participant.
  Other Names: PM+
  Arms: Stepped-care program (Step 1: DWM; Step 2: PM+)
Behavioral: Psychological First Aid (PFA) — PFA is a brief intervention consisting of providing basic information for peer support in times of emotional distress
  Other Names: PFA

SUMMARY:
Rationale: The COVID-19 pandemic has impacted the mental health of healthcare workers (HCWs). This study combines two low-intensity psychological interventions developed by the World Health Organization (Doing What Matters [DWM] and Problem Management Plus [PM+]) into a stepped-care program for HCWs.

Objective: The main objective is to evaluate the implementation and (cost-)effectiveness of the culturally and contextually adapted DWM/PM+ stepped-care programs amongst health care workers during the COVID-19 pandemic in terms of mental distress, resilience, wellbeing, health inequalities, and costs to health systems.

Study design: Phase 2 (intervention study): pragmatic implementation trial with a single-blinded, randomized, parallel-group design. Phase 3: qualitative process evaluation consisting of individual interviews and focus group discussions (FGDs).

Study population: Study phase 2: Health care workers with self-reported elevated psychological distress. Study phase 3: study participants with different trajectories through the trial (completers, non-completers, drop-outs, etc.), family members/close persons of participants, professionals, and facilitators of the DWM and PM+ intervention.

Intervention- study phase 2: All participants (in both the treatment and the comparison group) will receive Psychological First Aid (PFA) and care as usual (CAU). In addition to PFA and CAU, the treatment group will receive the stepped-care intervention (DWM with or without PM+) in addition to CAU. The stepped-care intervention consists of DWM (step 1) and conditionally PM+ (step 2) if participants still meet criteria for psychological distress (Kessler Psychological Distress scale (K10) >15.9) 1 month after having received DWM.

Main study parameters/endpoints: Phase 2: Screening for in- and exclusion criteria will be interviewer-administered, in-person or through (video) calls. Online assessments will take place at baseline, at 2 weeks after having received DWM, at 1 week and at 2 months after having received PM+. The main study parameter will be the decrease in symptoms of anxiety and depression from baseline to two-month follow-up, measured through the sum score of the Patient Health Questionnaire (PHQ-9) and General Anxiety Disorder-7 (GAD-7), i.e. the PHQ-Anxiety and Depression Score (PHQ-ADS). Phase 3: Through FGDs and interviews at the end of the study, the feasibility of scaling-up the implementation on the stepped-care DWM/PM+ intervention.

ELIGIBILITY:
Inclusion criteria:

* 18 years or older;
* Living in Madrid or Barcelona
* Having elevated levels of psychological distress (Kessler Psychological Distress Scale (K10) >15.9).
* Written/digital informed consent before entering the study.

Exclusion criteria:

* Having acute medical conditions (requiring hospitalization)
* Imminent suicide risk, or expressed acute needs, or protection risks that require immediate follow-up
* Having a severe mental disorder (e.g., psychotic disorders, substance-dependence)
* Having severe cognitive impairment (e.g., severe intellectual disability or dementia)
* Currently specialized psychological treatment (e.g., Eye movement desensitization and reprocessing, Cognitive behavioral therapy)
* In case of current psychotropic medication use, not being on a stable dose during the past 2 months being on an unstable dose for at least 2 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire Anxiety and Depression Scale (PHQ-ADS) | Change from baseline to 20 weeks
  The PHQ-ADS is a 16-item self-reported instrument that combines the nine-item Patient Health Questionnaire depression scale and seven-item Generalized Anxiety Disorder scale-as a composite measure of depression and anxiety. Respondents are asked how much each symptom has bothered them over the past 2 weeks, with response options of "not at all", "several days", "more than half the days", and "nearly every day", scored as 0, 1, 2, and 3. The scale can range from 0 to 48, with higher scores indicating higher levels of depression and anxiety symptomatology.

SECONDARY OUTCOMES:
Patient Health Questionnaire Anxiety and Depression Scale (PHQ-ADS) | Change: Baseline, 6 weeks, and 12 weeks
  The PHQ-ADS is a 16-item self-reported instrument that combines the nine-item Patient Health Questionnaire depression scale and seven-item Generalized Anxiety Disorder scale-as a composite measure of depression and anxiety. Respondents are asked how much each symptom has bothered them over the past 2 weeks, with response options of "not at all", "several days", "more than half the days", and "nearly every day", scored as 0, 1, 2, and 3. The scale can range from 0 to 48, with higher scores indicating higher levels of depression and anxiety symptomatology.
Patient Health Questionnaire (PHQ-9) | Change: Baseline, 6 weeks, 12 weeks, and 20 weeks
  The PHQ-9 is a 9-item self-reported instrument that measures depression symptoms. Respondents are asked how much each symptom has bothered them over the past 2 weeks, with response options of "not at all", "several days", "more than half the days", and "nearly every day", scored as 0, 1, 2, and 3. The scale can range from 0 to 27, with higher scores indicating higher levels of depression.
Generalized Anxiety Disorder (GAD-7) scale | Change: Baseline, 6 weeks, 12 weeks, and 20 weeks
  The GAD-7 is a 7-item self-reported instrument that measures anxiety symptoms. Respondents are asked how much each symptom has bothered them over the past 2 weeks, with response options of "not at all", "several days", "more than half the days", and "nearly every day", scored as 0, 1, 2, and 3. The scale can range from 0 to 21, with higher scores indicating higher levels of anxiety.
Posttraumatic Stress Disorder (PTSD) Checklist for Diagnostic and Statistical Manual of Mental Disorders (DSM-5) (PCL-5) - 8-item version | Change: Baseline, 6 weeks, 12 weeks, and 20 weeks
  The PCL-5 is a self-reported instrument that measures PTSD symptoms. Respondents are asked how much each symptom has bothered them over the past 4 weeks, with response options of "not at all", "a little bit", "moderately", "quite a bit", and "extremely". Items are rated on a 0-4 scale. The scale can range from 0 to 32 for the 8-item version, with higher scores indicating higher levels of PTSD symptoms.
EuroQol 5-dimensional descriptive system - 5-level version (EQ-5D-5L) | Change: Baseline, 6 weeks, 12 weeks, and 20 weeks
  The EQ-5D-5L measures quality of life and consists of two parts, the EQ-5D and the EQ VAS. Part 1, the EQ-5D, rates the level of impairment across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The labels for the 5L followed the format "no problems," "slight problems," "moderate problems," "severe problems," and "unable to"/"extreme problems" for all dimensions. For mobility, the description of "confined to bed" has been changed to "unable to walk about.". Part 2, the EQ-VAS, is a visual analogue scale. The endpoints of the scale are called 'The best health you can imagine' and 'The worst health you can imagine' and the current health status of that day needs to be indicated, after which the number checked on the scale also needs to be written down. Higher scores indicate worst qualitive of life.
Client Service Receipt Inventory (CSRI) - RESPOND adaptation | Change: Baseline, 6 weeks, 12 weeks, and 20 weeks
  The CSRI was developed for the collection of data on service utilization (e.g. use of health system, other services, time out of employment and other usual activities, need for informal care) and related characteristics of people with mental disorders, as the basis for calculating the costs of care for mental health cost-effectiveness research. The RESPOND-adapted version consists of a 13-item self-reported instrument that asks about the number and duration of contacts with healthcare professionals (physicians, mental health specialists, and nurses) in the past two months.
Stressor Reactivity | Change: Baseline, 6 weeks, 12 weeks, and 20 weeks
  Stressor reactivity (SR) is a proxy of resilience. SR scores are calculated based on the individual's association between stressor exposure, as measured by a checklist of daily hassles, and mental health, as measured by the Patient Health Questionnaire (PHQ-9) and the Generalised Anxiety Disorder (GAD-7) questionnaire. Residuals of individuals' regression lines are used to assess individual deviation from the normative SR (i.e., the SR in the RESPOND sample).

OTHER OUTCOMES:
Satisfaction with the intervention | 20 weeks
  Satisfaction with the intervention will be assessed through in depth interviews with participants, participants' relatives, and intervention deliverers
Positive Appraisal Style | Change: Baseline, 6 weeks, 12 weeks, and 20 weeks
  The Positive Appraisal Style Scale, content-focused (PASSc; in preparation), a 12-item self-report measure, to assess typical appraisal of stressors. Respondents are asked to rate the frequency of each item with the options 'never', 'sometimes', 'often', 'almost always', scored as 1, 2, 3, 4

CONTACTS AND LOCATIONS:
Overall Officials: José Luis Ayuso-Mateos, MD, PhD, Study Chair — Universidad Autonoma de Madrid; María Fe Bravo-Ortiz, MD, PhD, Principal Investigator — Hospital Universitario La Paz; Josep Maria Haro, MD, PhD, Principal Investigator — Parc Sanitari Sant Joan de Déu
Locations (2):
- Spain (2):
  - Parc Sanitari Sant Joan de Déu, Sant Boi de Llobregat, Barcelona
  - Hospital Universitario La Paz, Madrid

REFERENCES:
- [Derived] Mediavilla R, Garcia-Vazquez B, McGreevy KR, Underhill J, Bayon C, Bravo-Ortiz MF, Munoz-Sanjose A, Haro JM, Monistrol-Mula A, Nicaise P, Petri-Romao P, McDaid D, Park AL, Melchior M, Vuillermoz C, Turrini G, Compri B, Purgato M, Roos R, Witteveen AB, Sijbrandij M, Bryant RA, Fuhr D, Ayuso-Mateos JL. Beyond effectiveness in eHealth trials: Process evaluation of a stepped-care programme to support healthcare workers with psychological distress (RESPOND-HCWs). Digit Health. 2024 Oct 18;10:20552076241287678. doi: 10.1177/20552076241287678. eCollection 2024 Jan-Dec. PMID 39430699
- [Derived] Mediavilla R, Felez-Nobrega M, McGreevy KR, Monistrol-Mula A, Bravo-Ortiz MF, Bayon C, Gine-Vazquez I, Villaescusa R, Munoz-Sanjose A, Aguilar-Ortiz S, Figueiredo N, Nicaise P, Park AL, Petri-Romao P, Purgato M, Witteveen AB, Underhill J, Barbui C, Bryant R, Kalisch R, Lorant V, McDaid D, Melchior M, Sijbrandij M, Haro JM, Ayuso-Mateos JL; RESPOND Consortium. Effectiveness of a mental health stepped-care programme for healthcare workers with psychological distress in crisis settings: a multicentre randomised controlled trial. BMJ Ment Health. 2023 Jun;26(1):e300697. doi: 10.1136/bmjment-2023-300697. PMID 37263708
- [Derived] Mediavilla R, McGreevy KR, Felez-Nobrega M, Monistrol-Mula A, Bravo-Ortiz MF, Bayon C, Rodriguez-Vega B, Nicaise P, Delaire A, Sijbrandij M, Witteveen AB, Purgato M, Barbui C, Tedeschi F, Melchior M, van der Waerden J, McDaid D, Park AL, Kalisch R, Petri-Romao P, Underhill J, Bryant RA, Haro JM, Ayuso-Mateos JL; RESPOND Consortium. Effectiveness of a stepped-care programme of internet-based psychological interventions for healthcare workers with psychological distress: Study protocol for the RESPOND healthcare workers randomised controlled trial. Digit Health. 2022 Oct 5;8:20552076221129084. doi: 10.1177/20552076221129084. eCollection 2022 Jan-Dec. PMID 36211795